CLINICAL TRIAL: NCT01265121
Title: Sleep Apnea Syndrome on Acromegaly: Impact of the Treatment on the Carbohydrates Metabolism.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: InCor Heart Institute (Other)
Responsible Party: Felipe Henning Gaia Duarte, MD, Unit of Neuroendocrinology, discipline of endocrinology, University of São Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: FAPESP 2008/10045-3
Record Dates: First submitted 2010-12-13; First posted 2010-12-22 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-11

CONDITIONS: Acromegaly; Obstructive Sleep Apnea; Insulin Resistance
Keywords: Acromegaly; Insulin resistance; Euglycemic Clamp; Somatostatin analogues
MeSH Terms: conditions — Acromegaly; Sleep Apnea, Obstructive; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP treatment (Experimental): This acromegalic patients is going to have sleep apnea treated for 3 months with a with a continuous positive air pressure device (CPAP)
  Interventions: Device: Continuous positive air pressure device (CPAP)
- Nasal adhesive (Placebo Comparator): This acromegalic patients will be treated will an external nasal dilator adhesive intended to serve as a placebo treatment
  Interventions: Other: External nasal dilator adhesive

INTERVENTIONS:
Device: Continuous positive air pressure device (CPAP) — After titrating the air pressure during a polysomnography test, a CPAP device will be applied to the patient, during the night, for three months.
  Arms: CPAP treatment
Other: External nasal dilator adhesive — An external nasal dilator adhesive will be given to patients. They will be applied on the nose and will be used for three months aiming to serve as a placebo for snoring and sleep apnea.
  Other Names: Clear Passage (™) External nasal dilator adhesive
  Arms: Nasal adhesive

SUMMARY:
Sleep apnea is a common situation that affects up to 80% of acromegalic patients. This disease is linked to disturbance on the carbohydrate metabolism increasing the rates of diabetes. The objective of this trial is to assess (with the euglycemic hyperinsulinemic clamp) the impact of the treatment of sleep apnea, with a continuous positive air pressure device (CPAP), on the insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Acromegalic patients
* Moderate to severe sleep apnea
* Using somatostatin analogues at maximum dosage possible for at least 6 month

Exclusion Criteria:

* Unstable angina or high risk for stroke
* Hepatic or renal insufficiency
* Uncontrolled diabetes
* Seizures
* Steroids use
* Uncontrolled hormonal deficiencies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-04 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Assess the insulin resistance | At the beginning of the study and after 90 days.
  The insulin resistance, the target of this study, will be assessed by an index obtained during the euglucaemic hyperinsulinemic clamp (EHC). This index is derived from the amount of glucose delivered to the patient during a determined period of time. The (EHC) will be performed at the beginning of the study and 90 days after the intervention.

SECONDARY OUTCOMES:
Assess lipids profile and weight | At the beginning of the study and after 90 days.
  Lipids and weight will be assessed durind the study

CONTACTS AND LOCATIONS:
Overall Officials: Felipe HG Duarte, MD, Principal Investigator — Unit of neuroendocrinology, discipline of endocrinology, General Hospital of the University of São Paulo
Locations (1):
- General Hospital of the University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Amaro AC, Duarte FH, Jallad RS, Bronstein MD, Redline S, Lorenzi-Filho G. The use of nasal dilator strips as a placebo for trials evaluating continuous positive airway pressure. Clinics (Sao Paulo). 2012;67(5):469-74. doi: 10.6061/clinics/2012(05)11. PMID 22666791